CLINICAL TRIAL: NCT03827668
Title: A PHASE I, OPEN LABEL, FIXED SEQUENCE STUDY TO EVALUATE THE STEADY STATE PHARMACOKINETIC DRUG-DRUG INTERACTION BETWEEN PF-06650833 AND PF-06651600 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A DRUG-DRUG INTERACTION STUDY BETWEEN PF-06650833 AND PF-06651600 FOLLOWING MULTIPLE DOSES IN HEALTHY PARTICIPANTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7921028
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Drug-Drug Interaction
MeSH Terms: interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide; PF-06651600

STUDY DESIGN:
Intervention Model Description: This is a Phase I, open label, fixed sequence study. The study will consist of 2 periods in a single fixed sequence. In Period 1, participants will receive PF-06650833 once daily on Days 1-5 and PF-06650833 PK will be assessed for 24 hours following Day 5 dosing. Participants will be discharged on Day 6 after completion of study related activities. There will be a washout period of at least 7 days between last dosing in Period 1 and first dosing in Period 2. In Period 2, participants will receive PF-06651600 once daily alone on Days 1-7, and PF-06651600 once daily together with PF-06650833 once daily on Days 8-12. PF-06651600 PK will be assessed for 24 hours following Day 7 dosing, while PK for both PF-06651600 and PF-06650833 will be assessed for 24 hours following Day 12 dosing. Across both periods few additional pre-dose (trough) PK samples will be collected. Participants will remain in the unit up to Day 13 when they will be discharged after completion of study related activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): The study will have only one study group in a fixed-sequence type of design with two periods
  Interventions: Drug: PF-06650833 alone; Drug: PF-06651600 alone; Drug: PF-06650833 together with PF-06651600

INTERVENTIONS:
Drug: PF-06650833 alone — In Period 1, Days 1-5, participants will receive PF-06650833 once daily alone.
Drug: PF-06651600 alone — In Period 2, Days 1-7, participants will receive PF-06651600 once daily alone.
Drug: PF-06650833 together with PF-06651600 — In Period 2, Days 8-12, participants will receive PF-06650833 once daily together with PF-06650833 once daily.

SUMMARY:
The purpose of this study is to evaluate the potential pharmacokinetic (PK) drug-drug interaction (DDI) between PF-06650833 and PF-06651600 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD)
* Male and female participants who are healthy as determined by medical evaluation including medical history, physical examination, including blood pressure (BP) and pulse rate measurement, temperature, 12-lead ECG, and laboratory tests.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent as described in the protocol, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in the protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Known immunodeficiency disorder, including positive serology for human immunodeficiency virus (HIV) at screening, or a first degree relative with a hereditary immunodeficiency.
* Infection with hepatitis B or hepatitis C viruses according to protocol-specific testing algorithm.
* Participants with any of the protocol-listed acute or chronic infections or infection history.
* History of febrile illness within 5 days prior to the first dose of investigational product (in both Periods).
* History of any lymphoproliferative disorder such as Epstein Barr Virus (EBV) related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
* Participants have a known present or a history of malignancy other than a successfully treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* Benign ethnic (cyclic) neutropenia.
* Having received any live (attenuated) vaccines within 6 weeks prior to the first dose of investigational product.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* Previous administration of an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives (whichever is longer) preceding the first dose of investigational product used in this study.
* Known participation in a clinical trial of PF-06650833 or PF-06651600.
* A positive urine drug test at screening or admission.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* Participants with any of the protocol-listed abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary.
* Have evidence of untreated or inadequately treated active or latent Mycobacterium tuberculosis (TB) infection.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Use of tobacco/nicotine containing products in excess of 5 cigarettes/day.
* Have a history of major organ transplant or hematopoietic stem cell/marrow transplant. Skin grafts are allowed.
* Systemic therapy with any of the medications that are CYP3A4 inhibitors within 7 days or 5 half-lives (whichever is longer) or CYP3A4 inducers within 28 days or 5 half-lives (whichever is longer) prior to the first dose of the trial medication.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle Considerations criteria of the protocol.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
PF-06650833 Cmax | Fold-change from Period 1/Day 5 to Period 2/Day 12
  Maximum observed concentration (Cmax) derived from plasma
PF-06650833 AUCtau | Fold-change from Period 1/Day 5 to Period 2/Day 12
  Area under the plasma concentration-time profile derived from plasma from time 0 to time tau, the dosing interval (AUCtau), where tau=24 for QD dosing.
PF-06651600 Cmax | Fold-change from Period 2/Day 7 to Period 2/Day 12
  Maximum observed concentration (Cmax) derived from plasma
PF-06651600 AUCtau | Fold-change from Period 2/Day 7 to Period 2/Day 12
  Area under the plasma concentration-time profile derived from plasma from time 0 to time tau, the dosing interval (AUCtau), where tau=24 for QD dosing.

SECONDARY OUTCOMES:
Percentage of participants with treatment emergent adverse events | From screening until follow-up phone call that takes place 28-35 days after last study dose (total period of approximately 87 days)
Percentage of participants with clinical laboratory test results above/below certain threshold | At screening; Days -1, 6 in Period 1; and Days -1, 8, 9, 11, 13 in Period 2
Percentage of participants with vital signs above/below certain threshold | At screening; Days 1, 6 in Period 1; and Days 1, 8, 9, 12, 13 in Period 2
Percentage of participants with 12-lead electrocardiogram (ECG) results above/below certain threshold | At screening; Days 1, 6 in Period 1; and Days 1, 8, 9, 12, 13 in Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7921028